CLINICAL TRIAL: NCT02890212
Title: Double Blind, Placebo Controlled Pilot Study to Evaluate the Use of Selenium as an Augmentation Treatment for Sertraline Resistant Major Depression
Brief Title: Selenium as Augmentation Treatment for Sertraline Resistant Major Depression
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: due to COVID19 pandemic
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Teng Chei Tung, M. D. , Ph. D., University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Selen-2015
Record Dates: First submitted 2016-06-24; First posted 2016-09-07 (Estimated); Last update posted 2024-05-28 (Actual); Status verified 2024-05

CONDITIONS: Major Depression
Keywords: Major depression, selenium, placebo, sertraline
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- selenium (Experimental): subjects resistant to treatment of major depression with sertraline who were randomized and ingest selenium pills (400 microgram) during six weeks
  Interventions: Dietary Supplement: selenium supplementation
- placebo (Placebo Comparator): subjects resistant to treatment of major depression with sertraline who were randomized and ingest placebo pills
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: selenium supplementation — administration of selenium pills (400 micrograms) for randomized subjects
  Arms: selenium
Dietary Supplement: placebo — administration of placebo pills for randomized subjects
  Arms: placebo

SUMMARY:
The main goals of antidepressant treatments are to achieve remission of depressive episodes and prevent recurrences. However, clinical trials designed to approve antidepressants targets a response rate of at least 50%, which is considered partially effective. Therefore, there is a need for new treatment strategies, including augmentation with other substances such as lithium. This research aims to verify through a pilot study, the effect of selenium as an augmentation treatment for sertraline-resistant major depression. This clinical trial was designed to be a randomized, placebo-controlled, double-blind trial evaluating the effect of selenium or placebo in subjects diagnosed with major depression who have not responded to treatment with sertraline

DETAILED DESCRIPTION:
This research aims to verify in a pilot study the effect of selenium as an augmentation treatment for sertraline-resistant major depression and, as secondary endpoints, if the levels of selenium in patients with depressive episodes are different from individuals without depression. Thus, this clinical trial was intended to be a randomized double-blind placebo-controlled clinical trial evaluating the effect of selenium or placebo in patients diagnosed with major depression who have not responded to treatment with sertraline in appropriate dose and treatment duration. The initial sample will be comprised of patients with moderate or severe major depression, who will receive sertraline up to 200mg/day, for at least 8 weeks. A group of subjects without major depression will be selected as a control sample, which will be submitted to the same procedures of the included patients. It is estimated an initial sample of 90 patients with major depression (DSM-IV criteria), and about 30 patients resistant to treatment, which will be randomly divided into two groups (selenium and placebo). The control group sample is estimated to be 45 subjects.

For the diagnosis of major depression, it will be used the Structured Clinical Interview for DSM Axis I disorders (SCID Structured Clinical Interview for the DSM-IV Axis I disorders). To evaluate the outcome of treatment of the depressive symptoms, it will be used the Clinical Global Impression Scale and Patient Global Impression Scale (CGI and PGI), Hamilton Depression Rating Scale of 17 items for depression (HAM-D-17), Montgomery-Asberg Depression Rating Scale (MADRS) and SAFTEE- (brief structured interview assessing adverse events). The exclusion criteria include patients with any diagnosis of psychosis, bipolar disorder, personality disorder, any psychiatric condition that need hospitalization, severe risk of suicide, recent drug abuse or dependence, use of any polyvitamin substance, or any substance with known relevant psychopharmacological action, women with known or suspected pregnancy or breastfeeding, and people with unstable organic disease such as lupus erythematosus, uncontrolled diabetes mellitus, hypothyroidism and hyperthyroidism.

Participation is voluntary, and participants of both genders must be over the age of 18 years. After checking for exclusion and inclusion criteria (visit 0), the first phase of the study will start with the completion of the following laboratory tests: serum levels of selenium, electrocardiogram, hematology (hemoglobin, hematocrit, white blood cell count, platelet count), SGOT, SGPT, gammaGT, urea, creatinine, fasting glucose, TSH, free T4, T3, Na, K, total cholesterol + triglycerides fractions, urine analysis.

The second phase consists in the treatment of patients with depression with sertraline, which will receive initial dosage of 50 mg / day up to 200 mg or maximum tolerated dose, according to the investigator's decision, for at least 8 weeks. Patients considered resistant-sertraline (Hamilton-D-17> 7) will be invited to participate in the double-blind randomization phase to treatment groups with placebo or selenium (400 mcg / day). Sertraline will be maintained throughout the whole phase randomization. As the trial would be completed, participants will be referred to outpatient care in community health services. Initially the variables will be analyzed descriptively. In phase 1 Student's test will be used in order to compare the serum levels of selenium in both groups. At stage 2 for comparison of pre and post treatment with Sertraline it will be used the non-parametric McNemar test and in step 3, to determine the behavior of the groups during six weeks, it will be used analysis of variance with repeated measures.

ELIGIBILITY:
Inclusion Criteria:

1. of both genders
2. over the age of 18 years
3. in outpatient care
4. who meet the diagnostic criteria for major depression by the DSM-IV, confirmed by the application of structured interview SCID,
5. with scores higher than 17 on the Hamilton scale of 17 items for depression
6. who agree to participate voluntarily in the study, after full and unrestricted information about the study to be performed, as documented by signing the informed consent
7. Women of childbearing age need negative pregnancy test in the pre-assessment tests, and must use prevention of pregnancy during treatment.

Exclusion Criteria:

1. have a known sensitivity to sertraline or selenium
2. have psychiatric hospitalization indication, due to the presence of any psychiatric condition that would justify the hospitalization, including patients with severe risk of suicide.
3. have history of resistance to sertraline treatment, in clinical effective doses and for appropriate duration (at least 100 mg for at least 8 weeks).
4. have any psychosis (including diagnostic ICD10 F20-29, F06.0-06.2, F32.3 and F33.3), bipolar disorder or personality disorder
5. have received regular medication with psychotropic action the week prior to the trial inclusion
6. have received fluoxetine in the last four weeks prior to trial inclusion
7. have used any substance considered as a polyvitamin the week prior the inclusion
8. have received monoamine oxidase inhibitors 14 days prior to selection
9. show clinical diseases that require the use of medications that can interact with sertraline.
10. known or suspected pregnancy.
11. breast-feeding women.
12. Use of any drug that has known and relevant psychopharmacological action, despite not having preferential psychotropic drug use, unless it has been used with a stable dose for at least a month.
13. have dependency on any psychoactive substance in the last 12 months (except caffeine and tobacco).
14. Presence of an unstable disease that compromises the outcome (eg. Lupus Erythematosus, decompensated diabetes mellitus, cardiac insufficiency) that will determined clinically by the investigator.

For the control group, the same criteria of inclusion and exclusion above will be applied, except for the diagnosis of major depression by the DSM-IV and the scores of the Hamilton rating scale for depression.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2005-08 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Hamilton Depressive Rating Scale | 6 weeks

SECONDARY OUTCOMES:
Montgomery-Asberg Depression Rating Scale | 6 weeks
Clinical Global Impression Scale | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Teng C. Tung, M. D.,Ph. D., Principal Investigator — Hospital das Clinicas da Faculdade de Medicina da Universidade de São Paulo
Locations (1):
- Instituto de Psiquiatria - Hcfmusp, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ferrier IN. Treatment of major depression: is improvement enough? J Clin Psychiatry. 1999;60 Suppl 6:10-4. PMID 10235119
- [Background] McIntyre RS, O'Donovan C. The human cost of not achieving full remission in depression. Can J Psychiatry. 2004 Mar;49(3 Suppl 1):10S-16S. PMID 15147032
- [Background] Joffe RT, Levitt AJ. Relationship between antidepressant partial and nonresponse and subsequent response to antidepressant augmentation. J Affect Disord. 1999 Jan-Mar;52(1-3):257-9. doi: 10.1016/s0165-0327(97)00178-x. PMID 10357043
- [Background] Aronson R, Offman HJ, Joffe RT, Naylor CD. Triiodothyronine augmentation in the treatment of refractory depression. A meta-analysis. Arch Gen Psychiatry. 1996 Sep;53(9):842-8. doi: 10.1001/archpsyc.1996.01830090090013. PMID 8792761
- [Background] Rayman MP. The importance of selenium to human health. Lancet. 2000 Jul 15;356(9225):233-41. doi: 10.1016/S0140-6736(00)02490-9. PMID 10963212
- [Background] Hawkes WC, Hornbostel L. Effects of dietary selenium on mood in healthy men living in a metabolic research unit. Biol Psychiatry. 1996 Jan 15;39(2):121-8. doi: 10.1016/0006-3223(95)00085-2. PMID 8717610